# **HEALEY ALS Platform Trial - Regimen C CNM-Au8**

NCT04414345

**Document Date: 22 Jul 2022** 

# RGC REGIMEN-SPECIFIC STATISTICAL ANALYSIS PLAN (R-SAP)

**Master Protocol** Platform Trial for the Treatment of Amyotrophic Lateral

Sclerosis (ALS): A perpetual multi-center, multi-regimen,

clinical trial evaluating the safety and efficacy of investigational products for the treatment of ALS

**Regimen** RGC: CNM-Au8

Regimen Partner Clene Nanomedicine, Inc.

**Regulatory Sponsor** Merit E. Cudkowicz, MD

**Master Protocol Version** 4.0, 31 Aug 2020

**RSA Version** 5.0, 22 Nov 2021

Master SAP Version 1.0, 24 Jun 2020

**R-SAP Version** 3.0, 22 Jul 2022

#### SAP APPROVAL SIGNATURES

DocuSigned by Merit Cudkowicz

| Merit Cudkowicz | I approve this document<br> 07/22/2022 7:21:13 PM EDT | 07/22/2022 |
|---|---|---|
| Merit En Cudkowicz MD<br>Principal Investigator and | | Date |
| —DocuSigned by Sabrina Pag | anoni | |
| Sabrina Paganoni | I approve this document<br>07/22/2022 5:35:01 PM PDT | 07/22/2022 |
| Sabrina Paganoni MD P<br>Co-Principal Investigator | | Date |
| DocuSigned by Robert Glanz | zman | |
| | ove this document<br>/2022 5:06:10 PM PDT | 07/22/2022 |
| Robert Glanzman, MD F | GAAN<br>D386F-9400C<br>Iene Nanomedicine, Inc. | Date |

\_\_\_DocuSigned by Michael Hotchkin

Michael Hotchkin

07/22/2022

Michael Hotchkin Chief Development Officer, Clene Nanomedicine, Inc.

\_\_\_DocuSigned by Ben Saville

I approve this document 07/23/2022 | 12:54:46 PM EDT

07/23/2022

Date

Ben Saville PhD 50221BD2F3C9432B98632C6FEC7283AD Senior Statistical Scientist, Berry Consultants

DocuSigned by Eric A. Macklin

Eric A. Macklin

I approve this document 07/22/2022 | 7:06:09 PM EDT

07/22/2022

Eric A Macklin PhD 334DFC089673751 Study Biostatistician

Date

# SAP REVISION HISTORY

| Version | Date | Description of Changes |
|---|---|---|
| 1.0 | 17 Mar 2022 | Initial version |
| 2.0 | 09 May 2022 | Revision of Section 5.9 Survival to specify that both PAV-free survival and overall survival will be evaluated at both (i) the Week 24 Visit time point, and (ii) the last-participant-last-visit time point, and to specify that PAV-free survival to the Week 24 Visit time point is the primary analysis of survival in this analysis plan. |
| | | Revision of Section 6.5.2 CAFS to specify the following: |
| | | 1. A joint-rank analysis of PAV-free survival and SVC will be used as a supportive analysis for the secondary efficacy endpoint of SVC, |
| | | 2. The secondary endpoint joint-rank analyses will use multiple imputation to extend follow-up for participants who early terminate, withdraw consent, or are lost to follow-up as additional supportive analyses, |
| | | 3. The secondary joint-rank analyses will use time to death alone independent of any death equivalent as additional supportive analyses, and |
| | | 4. Primary inference from the joint-rank analyses will compare survival by time to death or death equivalent and will compare change in function to the last jointly observed time point. |
| 3.0 | 22 Jul 2022 | Revision of Section 4.2 Exploratory Endpoints to (i) identify serum creatinine, serum and CSF neurofilament light chain (NfL), and urinary p75[ECD] as exploratory biomarkers of neurodegeneration and neuromuscular degeneration, and (ii) include ALSAQ-40 domain scores and symptom index (SI) as exploratory endpoints. |
| | | Revision of Section 5.1 ALSFRS-R to specify details of the calculation of pre-baseline slope. |
| | | Revision of Section 5.5 Quantitative Voice Characteristics to include predicted vital capacity as an additional metric at the Baseline Visit. |
| | | Revision of Section 5.6 Biofluid Biomarkers of Neurodegeneration to specify assay techniques used to quantify serum creatinine, serum and CSF NfL, and urinary p75[ECD]. |

| Version | Date | Description of Changes |
|---|---|---|
| 3.0 (continued) | 22 Jul 2022<br>(continued) | Revision of Section 5.7 ALSAQ-40 to specify calculation of domain scores and to revise calculation of overall ALSAQ-40 SI. |
| | | Revision of Section 5.8 CNS-BFS to specify that the total score is referenced. |
| | | Revision of Section 5.9 Survival to specify that time at risk begins at each participant's Baseline Visit and to specify that the date of PAV initiation, where applicable, will be imputed as the fifteenth day of a month if not specified more precisely. |
| | | Revision of Section 6.1 Analysis Sets to add the Efficacy Common Mode of Administration (ECM) analysis set, to remove the restriction on protocol deviations that could be considered for exclusion from the Efficacy Per-protocol (EPP) analysis set must be classified as major protocol deviations, to specify the time point at which data is excluded from the EPP analysis set in the case of time-dependent exclusions, and to specify that data from placebo participants from other regimens would not be excluded from the EPP analysis set due to non-adherence to protocol-specified dosing. |
| | | Revision of Section 6.2 Baseline Characterization to include ALSAQ-40 domain scores and SI, urinary p75[ECD], and vital capacity predicted from quantitative voice characteristics. |
| | | Revision of Section 6.5.2 CAFS to clarify that the primary CAFS analysis is specified in the ALS Master Protocol Recommended Statistical Analysis, Design and Simulation Report and is an adjusted analysis, to provide code for an adjusted analysis, and to add three additional sets of CAFS analyses, one set that adjusts rank scores in linear models for time from ALS symptom onset, delta-FRS, baseline use of riluzole, and baseline use of edaravone, one set that adjusts for the same set of covariates plus baseline serum NfL level, and one that makes no adjustment. |
| | | Revision of Section 6.5.3 Repeated-measures Model to add a fixed term for treatment group (removing the shared-baseline assumption at the recommendation of the FDA) and to specify a separate supportive analysis that includes fixed terms for centered baseline serum NfL level, and centered baseline serum NfL level × visit interaction for analysis of clinical endpoints. |
| | | Revision of Section 6.5.4 Survival to include ECM as an additional analysis set, to include baseline age as an additional covariate in all adjusted models, and to specify an additional adjusted analysis that includes baseline serum NfL level. |

| Version | Date | Description of Changes |
|---|---|---|
| 3.0 (continued) | 22 Jul 2022<br>(continued) | Revision of Section 6.5.5 Random-slopes Model to add a fixed term for treatment group (removing the shared-baseline assumption) and to specify a separate supportive analysis that includes fixed terms for centered baseline serum NfL level, and centered baseline serum NfL level × study month interaction for analysis of clinical endpoints. |
| | | Revision of Section 6.5.7 Composite of ALSFRS-R, SVC, and ALSAQ-40 Slopes to specify that one analysis will adjust for years since ALS symptom onset, delta-FRS, baseline riluzole use, and baseline edaravone use, and an additional analysis will adjust for the same covariates plus baseline serum NfL level. |
| | | Revision of Section 6.5.8 HHD0 and HHD0 <sup>2</sup> to remove reference to the shared-baseline assumption of the repeated-measures mixed model of Section 6.5.3 and to specify a separate analysis that adds baseline serum NfL level as an additional covariate. |
| | | Revision of Section 6.5.9 Quantitative Voice Measures to remove reference to the shared-baseline assumption of the repeated-measures and random-slopes mixed models and to add a fixed term for treatment group (removing the shared-baseline assumption) and to specify a separate analysis that includes fixed terms for centered baseline serum NfL level, and centered baseline serum NfL level × B-spline interaction. |
| | | Revision of Section 6.5.10 Placebo Multiple Imputation to specify regression over sequential visits by the fully conditional specification method, to remove reference to the shared-baseline assumption of the repeated-measures mixed model of Section 6.5.3, and to specify a separate analysis that adds baseline serum NfL level as an additional covariate. |
| | | Revision of Section 6.5.13 Comparison of Controls across<br>Regimens to specify separate analyses that add baseline serum<br>NfL level as an additional covariate. |

#### **ABBREVIATIONS**

ALP Alkaline Phosphatase

ALS Amyotrophic Lateral Sclerosis

ALSAQ-40 Amyotrophic Lateral Sclerosis Assessment Questionnaire, 40-item version

ALSFRS-R Amyotrophic Lateral Sclerosis Functional Rating Scale, Revised

ALT Alanine Transaminase
AST Aspartate Transaminase

ATC WHODrug Anatomical, Therapeutic, and Chemical class

ATS American Thoracic Society

BLQ Below the Limit of Quantitation

BMI Body Mass Index

C-SSRS Columbia Suicide Severity Rating Scale

CAFS Combined Assessment of Function and Survival

CBC Complete Blood Count
CKD Chronic Kidney Disease
COVID-19 Coronavirus Disease 2019

CNS-BFS Center for Neurologic Study Bulbar Function Scale

CSF Cerebrospinal Fluid
CSR Clinical Study Report

CTCAE Common Terminology Criteria for Adverse Events

delta-FRS Pre-baseline Slope in ALSFRS-R

DAP Data Analysis Plan

DILI Drug-induced Liver Injury
DNA Deoxyribonucleic Acid

DRR Disease Rate Ratio

ECC Efficacy Concurrent Control

ECD Extra-cellular Domain

ECG Electrocardiography or Electrocardiogram

eGFR Estimated Glomerular Filtration Rate

EPP Efficacy Per-protocol
ERO Efficacy Regimen-only

ELISA Enzyme-linked Immunosorbent Assay

## ABBREVIATIONS (continued)

FAS Full Analysis Set

FVC Forced Vital Capacity
GLI Global Lung Initiative

hCG Human Chorionic Gonadotropin

HHD Hand-held Dynamometry

HLT MedDRA High Level Term

ICF Informed Consent Form

ITT Intention-to-treat Principle

M-SAP Master Statistical Analysis Plan

MDRD Modification of Diet in Renal Disease

MedDRA Medical Dictionary for Regulatory Activities

MP Master Protocol

MPRDR ALS Master Protocol Recommended Statistical Analysis, Design and

Simulation Report

NCI National Cancer Institute

NEALS Northeast ALS

NfL Neurofilament Light Chain
NIV Noninvasive Ventilation

OLE Open-label Extension

p75[ECD] Neurotrophin Receptor p75 Protein Extracellular Domain

PAV Permanent Assisted Ventilation

PD Pharmacodynamics
PK Pharmacokinetics

PT MedDRA Preferred Term

RBC Red Blood Cell

RDW RBC Distribution Width

RGC Regimen C (CNM-Au8, 30 mg/d and 60 mg/d)

RSA Regimen-specific Appendix

R-SAP Regimen-specific Statistical Analysis Plan

SAE Serious Adverse Event SAP Statistical Analysis Plan

## ABBREVIATIONS (continued)

SGOT Serum Glutamic Oxaloacetic Transaminase

SGPT Serum Glutamic Pyruvic Transaminase

SI Symptom Index

SoA Schedule of Activities

SOC MedDRA System Organ Class

SRO Safety Regimen-only

STF Safety and Tolerability Full

STN Safety and Tolerability Narrow

SVC Slow Vital Capacity

TBL Total Bilirubin

TEAE Treatment-emergent Adverse Event

TSH Thyroid Stimulating Hormone

ULN Upper Limit of Normal

WBC White Blood Cell

WHODrug World Health Organization Drug Dictionary Enhanced

# **Table of Contents**

| 1. | | overning Documents | |
|----|------|-----------------------------------------------------|----|
| 2. | Stı | tudy Design | 11 |
| | 2.1 | Overview | 11 |
| | 2.2 | Study Objectives | 12 |
| | | Study Population | |
| | | Participant Flow | |
| | | Regimen Allocation. | |
| | | Treatment Allocation. | |
| | | Treatment Administration | |
| | | Allocation Concealment | |
| | | RGC Schedule of Activities (SoA) | |
| 3. | | eneral Considerations for Data Analysis | |
| | | Statistical Software | |
| | | Summary Statistics | |
| | | Precision | |
| | | Transformations | |
| | | Multiplicity Adjustments | |
| | | Missing Data | |
| 4 | | tudy Endpoints | |
| т. | | Efficacy Endpoints | |
| | | Exploratory Endpoints | |
| | | Safety Endpoints | |
| _ | | leasurement Definitions | |
| э. | | ALSFRS-R | |
| | | SVC | |
| | | Home Spirometry | |
| | | HHD and Grip Strength | |
| | | Quantitative Voice Characteristics | |
| | | Biofluid Biomarkers of Neurodegeneration | |
| | | ALSAQ-40 | |
| | | CNS-BFS | |
| | | Survival | |
| | 5.10 | Pharmacokinetics of CNM-Au8 | |
| | 5.11 | King's ALS Clinical Staging System | 20 |
| | 5.12 | Hospitalization and Other Clinical Events | 21 |
| | 5.13 | Pharmacodynamic Biomarkers | |
| | 5.14 | Pharmacokinetics of Riluzole | |
| _ | 5.15 | Clinical Safety Laboratory Tests | |
| 6. | | tatistical Methodology | |
| | | Analysis Sets | |
| | | Baseline Characterization | |
| | | Primary Efficacy Analysis and Supportive Analyses | |
| | | Interim Analysis | |
| | | Secondary Efficacy Analyses | |
| | 6.5 | - | |
| | 6.5 | | |
| | 6.5 | 1 | |
| | 6.5 | | |
| | 6.5 | 1 | |
| | 6.5 | | |
| | | 5.7 Composite of ALSFRS-R, SVC, and ALSAQ-40 Slopes | |
| | 6.5 | | |
| | | 5.9 Quantitative Voice Measures | |
| | 6.5 | 5.10 Placebo Multiple Imputation | 32 |

| 6.5.11 | Additional Sensitivity Analyses of Primary and Key Secondary Outcomes | 32 |
|---|---|---|
| 6.5.12 | Subgroup Analyses | |
| 6.5.13 | Comparison of Controls across Regimens | |
| 6.5.14 | Pharmacokinetic Analyses of CNM-Au8 | 34 |
| 6.5.15 | Pharmacodynamic Biomarker Analyses | 34 |
| 6.5.16 | Pharmacokinetics of Riluzole | 34 |
| 6.6 Safe | ty Analyses | 34 |
| 6.6.1 | Treatment-emergent Adverse Events | 34 |
| 6.6.2 | Safety Labs | 35 |
| 6.6.3 | ECG Results | 35 |
| 6.6.4 | Vital Signs and Weight | 35 |
| 6.6.5 | Suicidality | 35 |
| 6.7 Othe | er Analyses | 35 |
| 6.7.1 | Participant Disposition | |
| 6.7.2 | Study Drug Compliance and Tolerance | 36 |
| 6.7.3 | Concomitant Medication Use | 36 |
| 6.7.4 | Medical History | 37 |
| 6.7.5 | Blindedness | 37 |
| 6.7.6 | Protocol Deviations | 37 |
| 6.7.7 | Impact of COVID-19 Pandemic | 37 |
| 7. Valida | tion | 37 |
| 7.1 Prim | nary Efficacy Analysis | 37 |
| | ondary, Exploratory, and Safety Analyses | |
| | ences | |

## 1. Governing Documents

This Regimen-specific Statistical Analysis Plan (R-SAP) for the CNM-Au8 regimen (RGC) specifies any modification from the default outcome measures, analysis samples, and planned analyses for the placebo-controlled period of the HEALEY ALS Platform Trial as specified in the Master SAP (M-SAP). The M-SAP and this R-SAP supplement the Master Protocol, the "ALS Master Protocol Recommended Statistical Analysis, Design and Simulation Report" (Appendix 1 to the Master Protocol), and the RGC Regimen-specific Appendix (RGC RSA). Please refer to the Master Protocol and the RGC RSA for details on the rationale for the study design, eligibility criteria, conduct of the trial, clinical assessments and schedule of assessments, definitions and reporting of adverse events, data management conventions, and regulatory oversight and compliance procedures. The "ALS Master Protocol Recommended Statistical Analysis, Design and Simulation Report" (MPRDR) and any regimen-specific deviations described in the RGC RSA, and this R-SAP are authoritative in defining the primary and interim analyses. In case of discrepancies between the RGC RSA and this R-SAP concerning use of shared placebos, this R-SAP is authoritative. In case of discrepancies between either SAP and the Master Protocol and the RGC RSA concerning matters of analysis other than the primary and interim analyses and use of shared placebos, the M-SAP and this R-SAP are authoritative. In case of discrepancies between the M-SAP and this R-SAP, this R-SAP is authoritative. On all matters not related to analysis, the Master Protocol and the RGC RSA are authoritative. The following table describes relationships among the relevant documents in adjudicating possible discrepancies with higher numbers indicating greater authority.

| Issues potentially requiring adjudication | Master<br>Protocol | RGC RSA | MPRDR | M-SAP | RGC<br>R-SAP |
|---|---|---|---|---|---|
| Use of shared placebos | 1 | 4 | 2 | 3 | 5 |
| Primary and interim analysis specifications not related to use of shared placebo | 1 | 5 | 4 | 2 | 3 |
| Statistical analysis specifications not related to use of shared placebo or primary and interim analyses | 1 | 3 | 2 | 4 | 5 |
| All matters not related to statistical analysis | 4 | 5 | 1 | 2 | 3 |

#### 2. Study Design

#### 2.1 Overview

The HEALEY ALS Platform Trial is a perpetual multi-center, multi-regimen clinical trial evaluating the safety and efficacy of investigational products for the treatment of ALS. RGC evaluates the safety and efficacy of CNM-Au8 administered orally at dosages of 30 mg/d and 60 mg/d vs. placebo. The RGC RSA describes the nature of the intervention and its mechanism of action, the mode and frequency of administration, additional eligibility criteria beyond those specified in the Master Protocol, additional enrollment procedures, and additions and modifications of safety and efficacy assessments relative to those outlined in the Master Protocol.


## 2.2 Study Objectives

Primary Efficacy Objective:

• To evaluate the efficacy of CNM-Au8 as compared to placebo on ALS disease progression.

Secondary Efficacy Objectives:

• To evaluate the effect of CNM-Au8 on selected secondary measures of disease progression, including survival.

Safety Objectives:

• To evaluate the safety of CNM-Au8 for ALS.

**Exploratory Efficacy Objectives:** 

- To evaluate the effect of CNM-Au8 on selected biomarkers and endpoints.
- To explore CNM-Au8 pharmacokinetics (PK) and pharmacodynamic (PD) effects.

# 2.3 Study Population

In addition to eligibility criteria specified in the Master Protocol, participants in RGC must not have a history of allergy to gold, gold salts, or colloidal gold preparations.

Participants will be recruited from approximately 60 centers located throughout the US that are part of the Northeast ALS (NEALS) Consortium.

## 2.4 Participant Flow

Participants in RGC follow the consenting, Master screening, regimen assignment, regimen-specific screening, randomization to active or placebo treatment, and follow-up procedures and timing described in the M-SAP. Detailed descriptions of study procedures and timing are specified in the Master Protocol and the RGC RSA.

## 2.5 Regimen Allocation

Participants in RGC are those determined eligible for Master Protocol-level inclusion and exclusion criteria and randomly assigned to RGC, stratified by use of: (i) riluzole, (ii) edaravone, (iii) both, or (iv) neither at the time of screening for the Master Protocol. Details of regimen assignment are described in the Platform Trial Regimen Assignment Plan.

#### 2.6 Treatment Allocation

Participants in RGC are randomly allocated in a 3:3:2 ratio to 30 mg/d CNM-Au8, 60 mg/d CNM-Au8, or placebo treatment based on a pre-specified permuted-block randomization schedule, stratified by use of (i) riluzole, (ii) edaravone, (iii) both, or (iv) neither at the time of screening for the Master Protocol.

#### 2.7 Treatment Administration

CNM-Au8 and placebo are supplied as pairs of bottles each containing 60 mL of liquid. Bottles of active study drug at the 30 mg/d dosage contain CNM-Au8 at a concentration of  $250 \text{ \mug/mL}$  (15 mg per bottle). Bottles of active study drug at the 60 mg/d dosage contain CNM-Au8 at a

concentration of  $500 \mu g/mL$  (30 mg per bottle). All formulations contain 32.8 mg sodium bicarbonate and  $60 \mu g/mL$  USP purified water.

A normal dosage is two (2) 60 mL bottles of study drug daily. If participants have difficulty tolerating study drug and with Site Investigator and Medical Monitor approval, participants may reduce the dosage to one (1) bottle daily. Participants who have down titrated may be rechallenged at full dosage with approval by the Site Investigator and Medical Monitor. Participants who cannot tolerate the rechallenge should remain at the dosage of one (1) bottle daily. Drug holidays (e.g., treatment-free periods) are not permitted.

The first dose of study drug should be administered while in the office/clinic on the day of the Baseline Visit after all visit assessments are complete. Additional details of treatment administration are described in the RGC RSA.

#### 2.8 Allocation Concealment

Allocation concealment is the same as described in the M-SAP. All formations of study drug are identical in appearance (size, shape, volume, and color) and smell.

# 2.9 RGC Schedule of Activities (SoA)

| | MP | RGC | Base- | Week | Week | Week | Week | Week | Week | Week | Final |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | Scrn <sup>1</sup> | Scrn <sup>2</sup> | line | 2 | 43 | 83 | 12 | 16 | 20 | 24 <sup>3</sup> | Call <sup>4</sup> |
| | Cln | Cln | Cln | Phn | Cln <sup>5</sup> | Cln <sup>5</sup> | Phn | Cln <sup>5</sup> | Phn | Cln | Phn |
| | -42d | -41d | Day | Day | Day | Day | Day | Day | Day | Day | 28d ±3 |
| Activity | to -1d | to 0d | 0 | 14±3 | 28±7 | 56±7 | 84±3 | 112±7 | 140±3 | 168±7 | ALD |
| Written Informed Consent <sup>6</sup> | X | X | | | | | | | | | |
| Inclusion/Exclusion Review <sup>7</sup> | X | X | | | | | | | | | |
| ALS & Medical History | X | | | | | | | | | | |
| Demographics | X | | | | | | | | | | |
| Physical Examination | X | | | | | | | | | | |
| Neurological Exam | X | | | | | | | | | | |
| Vital Signs <sup>8</sup> | X | | X | | X | X | | X | | X | |
| Slow Vital Capacity | $X^9$ | | X | | | C | | C | | X | |
| Home Spirometry | $X^9$ | | X | | | X | | X | | X | |
| Muscle Strength Assessment | | | X | | | С | | С | | X | |
| ALSFRS-R | X | | X | | X | X | X | X | X | X | |
| ALSAQ-40 | | | X | | | | | | | X | |
| CNS-BFS | | | X | | | X | | X | | X | |
| 12-Lead ECG | X | | | | | | | | | X | |
| Clinical Safety Labs <sup>10</sup> | X | | X | | X | X | | X | | X | |
| CNM-Au8 PK Samples <sup>11</sup> | | | X | | C | C | | | | X | |
| CNM-Au8 PD Samples <sup>11</sup> | | | X | | С | С | | | | X | |
| Biomarker Blood Collection <sup>11</sup> | | | X<br>X | | | C | | C | | X | |
| Biomarker Urine Collection <sup>11</sup> | | | | | | С | | С | | X | |
| DNA Collection <sup>12</sup> (optional) | | | X | | | | | | | | |
| CSF Collection (optional) | | | X | | | | | $C^{13}$ | | | |
| Concomitant Medication Review | X | X | X | X | X | X | X | X | X | X | |
| Adverse Event Review <sup>14</sup> | X | X | X | X | X | X | X | X | X | X | X |
| Suicidality C-SSRS | | | X | | X | X | | X | | X | |
| Install Smartphone Apps <sup>15</sup> | | | X | | | | | | | | |
| Smartphone Voice Recording <sup>16</sup> | | | X | | X | X | | X | | X | |
| Uninstall Smartphone App | | | | | | | | | | X | |
| Regimen Assignment | X | | | | | | | | | | |


| | MP<br>Scrn <sup>1</sup> | RGC<br>Scrn <sup>2</sup> | Base-<br>line | Week<br>2 | 43 | 83 | 12 | 16 | Week<br>20 | 24 <sup>3</sup> | Final Call <sup>4</sup> |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | Cln<br>-42d | Cln<br>-41d | Cln<br>Dav | Phn<br>Dav | Cln <sup>5</sup> Day | Cln <sup>5</sup> Day | Phn<br>Dav | Cln <sup>5</sup> Day | Phn<br>Dav | Cln<br>Dav | Phn 28d ±3 |
| Activity | to -1d | to 0d | 0 | 14±3 | 28±7 | 56±7 | 84±3 | 112±7 | 140±3 | 168±7 | ALD |
| Randomization within RGC | | | X | | | | | | | | |
| Administer/Dispense Study Drug | | | $X^{17}$ | | | X | | X | | | |
| Drug Accountability/Compliance | | | | $X^{18}$ | X | X | $X^{18}$ | X | $X^{18}$ | X | |
| Exit Questionnaire | | | | | | | | | | X | |
| Vital Status | | | | | | | | | | $X^{19}$ | |

Abbreviations: ALD = after last dose, ALS = amyotrophic lateral sclerosis, ALSAQ-40 = ALS Assessment Questionnaire, ALSFRS-R = ALS Functional Rating Scale Revised, BP = blood pressure, C = completed only if the visit is conducted in-clinic, CBC = complete blood count, Cln = Clinic visit, CNS-BFS = Center for Neurologic Study Bulbar Function Scale, CSF = cerebrospinal fluid, C-SSRS = Columbia-Suicide Severity Rating Scale, d = day, DNA = deoxyribonucleic acid, ECG = electrocardiogram, LFTs = liver function tests, MP = Master Protocol, PD = pharmacodynamic, Phn = Phone visit, RGC = the CNM-Au8 regimen, Scrn = Screening Visit.


<sup>&</sup>lt;sup>1</sup> Master Protocol (MP) screening procedures must be completed between 42 days and 1 day prior to the Baseline Visit.

<sup>&</sup>lt;sup>2</sup> RGC regimen-specific screening procedures must be completed no more than 41 days prior to the Baseline Visit. RGC regimen-specific screening procedures may be completed on the same day as the Baseline Visit.

<sup>&</sup>lt;sup>3</sup> Participants should be instructed to hold the morning dose of study drug on the day of the Week 4, 8, and 24 study visits. Study drug should not be taken until after study visit procedures are complete.

<sup>&</sup>lt;sup>4</sup> Participants who are participating into the Open-label Extension (OLE) at the time scheduled for the Follow-up Safety Call will not complete a Follow-up Safety Call. Participants who continue into the OLE and then terminate prior to the time scheduled for the Follow-up Safety Call should be asked to complete a Follow-Up Safety Call.

<sup>&</sup>lt;sup>5</sup> The Week 4, 8, and 16 visits may be conducted via telemedicine (or via phone if telemedicine is not available) with remote services instead of in-clinic if this is needed to protect the safety of the participant due to a pandemic, or other reason. If a planned in-clinic visit is conducted via telemedicine (or via phone if telemedicine is not available) with remote services, only selected procedures will be performed: ALSFRS-R, home spirometry (Weeks 8 and 16 only), Center for Neurologic Study Bulbar Function Scale (CNS-BFS, Weeks 8 and 16 only), voice recording, adverse event review, Columbia Suicide Severity Rating Scale, concomitant medications, study drug accountability/compliance, and administer/dispense study drug. Additionally, selected vital signs (systolic and diastolic pressure, respiratory rate, heart rate, and temperature) and clinical safety labs will be performed by a home health agency.

<sup>&</sup>lt;sup>6</sup> During the Master Protocol Screening Visit, participants will be consented using the Master Protocol informed consent form (ICF). After a participant is randomly assigned to RGC, he or she will be consented a second time using the RGC ICF.

- <sup>7</sup> At the MP Screening Visit, participants will have MP inclusion and exclusion criteria assessed. At the RGC Screening Visit, participants will have regimen-specific inclusion and exclusion criteria assessed.
- <sup>8</sup> At all visits, whether conducted in-clinic or via telemedicine (or via phone if telemedicine is not available), vital signs include systolic and diastolic blood pressure, heart rate, respiratory rate, and temperature. At all in-clinic visits, vital signs include weight. At the MP Screening Visit only, vital signs include height measured in cm.
- <sup>9</sup> If required due to pandemic-related restrictions, forced vital capacity (FVC) performed by a Pulmonary Function Laboratory evaluator or with a study-approved home spirometer or sustained phonation using a study-approved method may be used for eligibility (Master Protocol Screening ONLY).
- <sup>10</sup> Clinical safety labs include hematology (CBC with differential), complete chemistry panel, liver function tests, thyroid function, and urinalysis. Serum pregnancy testing will occur in women of child-bearing potential at the Master Protocol Screening Visit and as necessary during participation. Pregnancy testing is only repeated as applicable if there is a concern for pregnancy.
- <sup>11</sup> Whole blood samples for CNM-Au8 PK, plasma samples for riluzole PK, and whole blood, plasma, and urine samples for PD biomarkers should be obtained prior to the first daily dose of study drug at each applicable clinic visit. The time of the most recent dose of study drug, the most recent meal prior to sampling, and the time of sample collection should be reported. Whole blood and urine will be collected only at the Baseline and Week 24/Early Termination visits.
- <sup>12</sup> If the participant consents to DNA sample collection but a DNA sample is not obtained at the Baseline Visit or if that sample is not usable, a DNA sample can be collected after the Baseline Visit.
- <sup>13</sup> If the participant consents to CSF sample collection but a CSF sample is not obtained at the Week 16 Visit, a CSF sample can be collected at the Week 24 Visit.
- <sup>14</sup> Adverse events that occur after signing the RGC ICF will be recorded.
- <sup>15</sup> Two smartphone apps should be installed on the participant's phone, one to collect home spirometry and one to collect voice recordings.
- <sup>16</sup> In addition to study visits specified in the SoA for collection of voice recordings, participants should complete twice weekly voice recordings at home. During weeks when a participant completes a voice recording in-clinic, he or she should only complete one other voice recording at home.
- <sup>17</sup> Administer first dose of study drug only after Baseline Visit procedures are completed. Participants should take the first dose of study drug while in the office/clinic on the day of the Baseline visit.
- <sup>18</sup> Drug accountability will not be done at phone visits. A drug compliance check-in must be held during phone visits to ensure participant is taking drug per dose regimen and to note any report of missed doses.
- <sup>19</sup> Vital status, a determination of date of death or death equivalent or date last known alive, will be made for each randomized participant at the end of their double-blind follow-up (generally the Week 24 Visit as indicated) and again, if previously alive, after the end of double-blind follow-

up of all participants randomized to RGC. Vital status may also be ascertained at later time points by using publicly available data sources.

#### 3. General Considerations for Data Analysis

#### 3.1 Statistical Software

Statistical software use for analyses is the same as described in the M-SAP.

## 3.2 Summary Statistics

Data summaries are the same as described in the M-SAP.

### 3.3 Precision

Precision of reported results is the same as described in the M-SAP.

#### 3.4 Transformations

Data transformations are the same as described in the M-SAP.

## 3.5 Multiplicity Adjustments

Handling of multiplicity adjustments is the same as described in the M-SAP with the addition that the primary contrast for any given analysis will be between all active arm participants (i.e., both 30 mg/d and 60 mg/d dosage groups) vs. placebo participants. Comparisons between the two dosage groups and between each dosage group and placebo will be exploratory.

#### 3.6 Missing Data

Handling of missing data is the same as described in the M-SAP. Clinic-based assessments that are missing due to COVID-19 restrictions or disruptions are considered missing at random.

#### 4. Study Endpoints

## 4.1 Efficacy Endpoints

The primary endpoint is the same as described in the M-SAP. ALSFRS-R total score is considered the primary efficacy endpoint as described in the M-SAP. Combined assessment of function and survival (CAFS), slow vital capacity (SVC) change, and survival (time to death or death equivalent) are considered key secondary efficacy endpoints in RGC.

## 4.2 Exploratory Endpoints

The following categories of exploratory endpoints will be evaluated:

- Change in ALSFRS-R domain scores,
- Change in strength: hand-held dynamometry (HHD) global percentage, HHD upper extremity percentage, HHD lower extremity percentages, HHD0, and HHD0<sup>2</sup>,


- Change in quantitative voice characteristics as measured by Aural Analytics: maximum phonation time, pause rate, breathy vocal quality, pitch instability, regulation of voicing, articulatory precision, speaking rate, articulation rate, and monotonicity,
- Change in biofluid biomarkers of neurodegeneration and neuromuscular degeneration: serum creatinine, serum and cerebrospinal fluid (CSF) neurofilament light chain (NfL), and urinary neurotrophin receptor p75 protein extracellular domain (p75[ECD]) normalized to urinary creatinine,
- Change in patient-reported outcomes: ALSAQ-40 physical mobility, independence in activities of daily living, eating and drinking, communications, and emotional reactions domain scores and ALSAQ-40 symptom index, CNS-BFS total score,
- Change in plasma and whole blood concentrations of CNM-Au8,
- Change in CNM-Au8 PD biomarkers,
- Change in respiratory function as assessed by home spirometry,
- Time to clinical events:
  - o First hospitalization due to a serious adverse event (SAE),
  - o First hospitalization due to an ALS-related SAE,
  - o First use of assisted ventilation,
  - o First placement of a feeding tube,
  - o First time reaching King's stage 4a or 4b,
  - First instance of any of the following events: feeding tube placement, tracheostomy, initiation of permanent assisted ventilation (PAV), or death,
  - o First instance of any of the following events: hospitalization for an SAE, feeding tube placement, tracheostomy, initiation of PAV, or death.
- Time to first occurrence of a  $\geq$  6-point decline in ALSFRS-R total score
- A composite of the standardized slope estimates for rate of change in ALSFRS-R total score, SVC percent-predicted, and ALSAQ-40 total score.

## 4.3 Safety Endpoints

In addition to the safety endpoints described in the M-SAP, the following RGC regimen-specific safety endpoint will be evaluated:

- Safety lab alerts: Proportion of participants with ALT >3x upper limit of normal (ULN), AST >3x ULN, creatinine >1.5x level at the Baseline Visit, and platelet count <75,000/mm<sup>3</sup>, and
- Pharmacokinetics of riluzole.

#### 5. Measurement Definitions

#### 5.1 ALSFRS-R

The definitions of ALSFRS-R scores are the same as described in the M-SAP. Pre-baseline slope in ALSFRS-R (delta-FRS) is defined as 48 minus the baseline ALSFRS-R total score then divided by the number of months from onset of symptomatic weakness to the Baseline Visit. The number of months will be calculated as the difference in days from onset of symptomatic weakness to the Baseline Visit multiplied by 12 / 365.25. The date of onset of symptomatic weakness will be imputed as the fifteenth day of a month if not specified more precisely.

ALSFRS-R domain scores are exploratory measures of the primary efficacy endpoint ALSFRS-R total score.

Time to first occurrence of a  $\geq$  6-point decline in ALSFRS-R total score is a composite endpoint with death or death equivalent, whichever occurs first, and will be censored at the last date at which an ALSFRS-R assessment was performed up to the end of the Week 24 Visit window.

#### **5.2** SVC

The derivation of SVC percent-predicted of normal is the same as described in the M-SAP with age calculated as number of days from date of birth to the date of a given SVC assessment divided by 365.25 and with the following correspondence between self-identified race and race defined by Global Lung Initiative (GLI) classification:

| Self-identified Race | GLI-defined Race |
|-------------------------------------------|------------------|
| American Indian or Alaska Native | Mixed/Other |
| Asian | South East Asian |
| Black or African American | African American |
| Native Hawaiian or Other Pacific Islander | Mixed/Other |
| White | Caucasian |
| Unknown | Caucasian |
| Not reported | Caucasian |
| More than one race indicated | Mixed/Other |

# **5.3** Home Spirometry

Home spirometry assesses FVC remotely using a smartphone app (ZEPHYRx, Albany, NY) and a handheld spirometer (Spirobank Smart, Medical International Research, Rome, Italy). Coordinators guide participants through 3 to 8 maneuvers with live-video coaching using the ZEPHYRx platform. Flow loops are classified for acceptability and repeatability using American Thoracic Society (ATS) criteria and are manually reviewed by the NEALS Outcomes Center (Barrow Neurological Institute, Phoenix, AZ). The maximum FVC accepted by the NEALS Outcomes Center is converted to percent of predicted normal using GLI norms based on sex, age at time of assessment, height at time of screening, and race. Age is calculated as number of days from date of birth to the date of a given home spirometry assessment divided by 365.25. Higher values indicate greater respiratory function.


## 5.4 HHD and Grip Strength

The derivation of HHD upper and lower extremity scores and HHD0 are the same as described in the M-SAP with the revision that HHD0 is a composite endpoint with death or death equivalent.

A second HHD time-to-event endpoint is defined as the time from the Baseline Visit to the second post-baseline occurrence of a muscle with a strength recording of 0 among those muscles that were non-zero at baseline, or time to death or death equivalent, whichever occurs first (HHD0<sup>2</sup>).

Time at risk for HHD0 and HHD0<sup>2</sup> will be censored at the last date at which an HHD assessment was performed up to the end of the Week 24 Visit window.

HHD lower extremity average percentage, HHD upper extremity average percentage, HHD global average percentage, HHD0, and HHD0<sup>2</sup> are exploratory measures.

## 5.5 Quantitative Voice Characteristics

Voice samples will be collected using the Aural Analytics app installed on either an Android or iOS-based smartphone. At each assessment, participants perform a set of speaking tasks: reading 5 prespecified sentences, reading 5 sentences chosen at random from a large sentence bank, repeating a consonant-vowel sequence, producing a sustained phonation, and counting on a single breath. Speech analysis will be performed by Aural Analytics to derive the following quantitative voice characteristics: maximum phonation time, pause rate, breathy vocal quality, pitch instability, regulation of voicing, articulatory precision, speaking rate, articulation rate, and monotonicity. Aural Analytics will use data on quantitative voice characteristics and participant age, sex, race, height, and weight to derive a prediction of vital capacity at the Baseline Visit.

## 5.6 Biofluid Biomarkers of Neurodegeneration

Biofluid biomarkers of neurodegeneration, including biomarkers of neuromuscular dysfunction, will be assayed. These will include serum creatinine, serum and CSF neurofilament light chain (NfL), and urinary p75[ECD]. Serum creatinine will be assayed by the kinetic Jaffe method (test 001370, Labcorp, Burlington, NC). NfL will be assayed by single-molecule array (Simoa; Quanterix, Billerica, MA). Urinary p75[ECD] will be assayed by sandwich enzyme-linked immunoassay (Rogers lab, Flinders Univ, Adelaide, Australia) and normalized to urinary creatinine. Levels of serum and CSF NfL and urinary p75[ECD] that are reported to be below the limit of quantitation will be imputed at the limit of quantitation. Levels of serum and CSF NfL will be log-transformed in all analyses.

#### 5.7 ALSAO-40

The description of the ALSAQ-40 instrument and item-level scores are the same as described in the M-SAP. Each of the five domains will be scored as the mean of all domain-specific items multiplied by 25 (range 0 to 100). An overall symptom index (SI) will be scored as the mean of the five domain scores. A domain score will be missing if more than 20% of the items are missing; otherwise, item non-response will be mean-imputed from other completed items from the same assessment. The ALSAQ-40 SI will be missing if any domain scores are missing. Higher scores indicate worse quality of life.


#### 5.8 CNS-BFS

The definition of CNS-BFS total score is the same as described in the M-SAP.

#### 5.9 Survival

The primary definition of survival time is the same as described in the M-SAP with the clarification that PAV is defined as more than 22 hours per day of noninvasive or invasive mechanical ventilation for more than seven consecutive days. The date of PAV initiation, where applicable, will be imputed as the fifteenth day of a month if not specified more precisely. A secondary survival endpoint of death alone, independent of any death equivalent, is also defined.

Time at risk for the composite endpoint of death or death equivalent and time at risk for the endpoint of death alone will be measured from each participant's Baseline Visit. Time at risk will be censored at two time points: (1) at the Week 24 Visit as defined in the M-SAP, and (2) at a subsequent assessment of death or death equivalent scheduled approximately at the end of placebo-controlled follow-up of the last RGC participant, with the latter effectively a comparison of either no-treatment or 24-week delayed treatment (for those participants who enter the openlabel extension). The primary analysis of survival will evaluate PAV-free survival to the Week 24 Visit time point.

#### 5.10 Pharmacokinetics of CNM-Au8

Whole blood and plasma samples collected at the Baseline and Week 24 visits will be analyzed to quantify the concentration of CNM-Au8. Details of the CNM-Au8 assay technique and analysis plan will be specified in a separate PK analysis plan. This plan will be finalized prior to database lock.

## 5.11 King's ALS Clinical Staging System

The King's ALS Clinical Staging System (Roche et al. 2012) is a 4-level ordinal scale with the first three levels indicating the number (1, 2, or 3) of distinct central nervous system regions (bulbar, upper limb, and lower limb) with neuromuscular dysfunction and levels 4a and 4b indicating nutritional or respiratory failure secondary to ALS, respectively.

Participants will be classified to King's stage 1, 2, 3, 4a, or 4b based on scores from ALSFRS-R assessments according to a published derivation (Balendra et al. 2014). Bulbar involvement is defined as a score less than 4 on any of the ALSFRS-R questions in the bulbar domain (questions 1, 2, and 3). Upper limb involvement is defined as a score less than 4 on either of the ALSFRS-R questions related to hand function (questions 4 and 5A). Lower limb involvement is defined as a score less than 4 on the ALSFRS-R question about walking (question 8). Nutritional failure is defined as responding that the participant uses gastrostomy for greater than 50% of their nutrition. Respiratory failure is defined as a score of 0 on the ALSFRS-R question addressing dyspnea (question 10 or R-1) or a score less than 4 on the ALSFRS-R question about use of mechanical ventilation (question 12 or R-3). Participants without evidence by ALSFRS-R scores of involvement of any of the three central nervous system regions will be scored as King's stage 1 due to their confirmed diagnosis with ALS. Participants may meet criteria for both King's stage 4a and 4b.


## 5.12 Hospitalization and Other Clinical Events

Times to the following clinically relevant events are defined:

- Time to first hospitalization due to a serious adverse event (SAE),
- Time to first hospitalization due to an ALS-related SAE,
- Time to first use of assisted ventilation,
- Time to first placement of a feeding tube,
- Time to King's stage 4a or 4b,
- Time to first instance of feeding tube placement, tracheostomy, initiation of PAV, or death, and
- Time to first instance of hospitalization for an SAE, feeding tube placement, tracheostomy, initiation of PAV, or death.

Time at risk for each event will be measured from each participant's Baseline Visit. Time to first hospitalization excludes hospitalizations for elective procedures. ALS-related SAEs are those indicated as related to ALS disease progression by the site investigator. Participants will be excluded from respective analysis (as applicable) if: (i) they are already using assisted ventilation or have a feeding tube at the time of the Baseline Visit, (ii) they have answered Question 5B on the ALSFRS-R at the Baseline visit, or (iii) have scored 0 points on Question 10 or less than 4 points on Question 12 of the ALSFRS-R at the Baseline visit. Death or death equivalent will be considered an outcome for each of the events listed, forming a composite endpoint.

Time at risk for these events will be censored at the Week 24 Visit, if completed, the date of consent withdrawal, if withdrawn, or the last date at which the status of each endpoint is known prior to the end of the Week 24 Visit window for participants lost to follow-up. Time to King's stage 4a or 4b is interval censored between ALSFRS-R assessments.

#### 5.13 Pharmacodynamic Biomarkers

Whole blood and urine PD samples collected at the Baseline and Week 24 visits and plasma PD samples collected at the Baseline, Week 4, Week 8, and Week 24 visits will be analyzed according to a separate PD analysis plan. The PD analysis plan will be finalized prior to database lock.

#### 5.14 Pharmacokinetics of Riluzole

Plasma samples collected at the Baseline, Week 4, and Week 8 visits from the first forty (40) RGC participants taking riluzole who reach the Week 8 visit plus plasma samples collected at the Baseline Visit from an additional ten (10) RGC participants not taking riluzole will be analyzed to quantify riluzole concentration by high-performance liquid chromatography mass spectroscopy (LC/MS/MS) [Covance, Method ID: M10125, Study Number 8454-985].

#### **5.15** Clinical Safety Laboratory Tests

Clinical safety labs include hematology, blood chemistry panel, liver function tests, thyroid function, urinalysis, and pregnancy testing in women of childbearing potential as specified in Section 9.1.2 Clinical Safety Laboratory Tests of the Master Protocol:

- Hematology: hematocrit, hemoglobin, platelet count, red blood cell (RBC) count, mean
  corpuscular volume, mean corpuscular hemoglobin, mean corpuscular hemoglobin
  concentration, RBC distribution width (RDW), RBC morphology, white blood cell (WBC)
  count, and counts and percentages of basophils, eosinophils, lymphocytes, monocytes, and
  neutrophils;
- Blood chemistry panel: bicarbonate, chloride, potassium, sodium, calcium, magnesium, phosphate, blood urea nitrogen, creatinine, estimated glomerular filtration rate (eGFR) calculated using the Modification of Diet in Renal Disease (MDRD) four-variable equation, creatinine clearance calculated using the Cockcroft-Gault equation, and glucose;
- Liver function tests: alanine aminotransferase (ALT [SGPT]), aspartate aminotransferase (AST [SGOT]), alkaline phosphatase (ALP), albumin, total protein, total bilirubin (TBL);
- Thyroid function tests: thyroid-stimulating hormone (TSH);
- Urinalysis: clarity, color, specific gravity, pH, microalbumin, protein, glucose, ketones, bilirubin, urobilinogen, nitrite, leukocyte esterase, and blood; and
- Pregnancy: qualitative and quantitative serum human chorionic gonadotropin (hCG).

Clinical safety labs will also include derived measures of potential drug-induced liver injury (DILI), including those that potentially meet the Hy's law criteria, as distinct safety lab outcomes.

Three potential DILI criteria will be defined:

- ALT or AST >3x ULN with TBL >1.5x ULN
- AST or ALT >3x ULN with TBL >2x ULN
- AST or ALT >3x ULN with TBL >2x ULN and ALP <2x ULN (potential Hy's Law cases) where ULN is upper level of normal and all levels are measured on the same day.

#### 6. Statistical Methodology

#### 6.1 Analysis Sets

The ITT analysis set is henceforth referred to as the Full Analysis Set (FAS) and defined as follows:

• Full Analysis Set (FAS): Participants who were randomized within RGC plus placebo participants from specified regimens, classified according to their randomized treatment assignment. Observations made after premature permanent discontinuation of study drug are included in this sample, should such participants remain on study. Observations completed after regimen data lock are excluded. Participants determined to not meet ALS diagnostic criteria are excluded.

The definition of the STF analysis set is revised as follows:

• Safety Full (STF) Set: Participants who initiated treatment within RGC plus placebo participants from specified regimens who are not known to be ineligible for RGC and who initiated treatment in their respective regimen, classified according to the treatment they

actually received. Observations made after premature permanent discontinuation of study drug are included in this sample, should such participants remain on study. Observations completed after regimen data lock are excluded.

An analysis set restricting shared placebo participants to those regimens in which study drug is administered by the same route as RGC is defined as follows:

• Efficacy Common Mode of Administration (ECM) Set: The subset of participants in the FAS analysis set who are in regimens in which study drug is administered by the same route as RGC (oral administration).

The definitions of the ECC, ERO, STN, and SRO analysis sets are the same as described in the M-SAP with reference to the ITT analysis set now referencing the FAS analysis set. The following analysis set is specific to RGC:

• Efficacy Per-protocol (EPP) Set: The subset of participants in the FAS analysis set who initiated study treatment and who were not involved in protocol deviations that affected the scientific integrity of the trial as documented prior to data lock, classified according to the treatment they actually received. Inclusion or exclusion from the EPP analysis set of any participant for whom treatment assignment was unblinded prior to data lock will be governed by the prespecified criteria above. If a participant's data is truncated for inclusion in the EPP analysis set due to non-adherence to protocol-specified dosing, clinical events observed up to 28 days after the censoring event will be included in the EPP analysis set. For all other events leading to truncation of a participant's data, no events beyond that date will be included. Data from placebo participants shared from other regimens will not be truncated due to non-adherence to protocol-specified dosing.

Applicable analysis sets (FAS, ECM, EPP, STF, and STN) will include shared placebo participants from regimens A, B, and D. Data from shared placebo participants will include visits and events that occurred on or before the date of the final placebo-controlled period follow-up of an RGA, RGB, or RGC participant. As only concurrently enrolling regimens are contributing to efficacy analyses, the FAS and ECC analysis sets are synonymous and only the FAS analysis set will be referenced. As regimen A is administered by subcutaneous injection and regimens B and D are administered orally, only regimens B and D will contribute shared placebo participants for the ECM and STN analysis sets.

#### **6.2** Baseline Characterization

The baseline characteristics summarized for participants randomized within RGC are the same as specified in the M-SAP with the addition of ALSAQ-40 domain scores and SI, CNS-BFS total score, King's stage, weight, body mass index (BMI), serum urate concentration, serum creatinine concentration, serum NfL concentration, urinary p75[ECD], and vital capacity predicted from quantitative voice characteristics.

## 6.3 Primary Efficacy Analysis and Supportive Analyses

The primary analysis for RGC is a Bayesian shared-parameter, repeated-measures model of ALSFRS-R that accounts for loss of follow-up due to mortality. Details of the model, including documentation of operating characteristics under a range of scenarios, are provided in the "ALS Master Protocol Recommended Statistical Analysis, Design and Simulation Report" (Appendix 1 to the Master Protocol). The Bayesian shared-parameter, repeated-measures model will be

applied to the FAS analysis set as the primary analysis, to the ECM and ERO analysis sets as sensitivity analyses, and to the EPP analysis set as a supportive analysis.

The estimand of the primary analysis is the relative rate of disease progression (the "disease rate ratio" or DRR) of the two active treatment groups relative to placebo in the FAS population under an assumption that active treatment slows mean time to death or death equivalent by the same proportion as treatment slows the mean rate of functional progression as measured by change in ALSFRS-R total score over time. The estimand is defined by the following attributes:

- Treatment: CNM-Au8 administered orally at dosages of 30 mg/d and 60 mg/d vs. placebo.
- Population: FAS population as defined in Section 6.1.
- Variables: time to death or death equivalent and rate of change in ALSFRS-R total score from baseline to the Week 24 Visit.
- Intercurrent event 1: treatment discontinuation due to death: no ALSFRS-R data from participants who reach the death or death equivalent endpoint are included in the analysis; instead, death or death equivalent are handled by a mortality component within the model, composite variable strategy approach.
- Intercurrent event 2: treatment discontinuation not due to death: handled via treatment policy approach, all data will be used including data collected during the placebo-controlled period after treatment discontinuation regardless of concomitant medication, for those participants who have not been censored due to mortality. Missing data post-treatment will not be imputed, handled via missing at random assumption.
- Population-level summary: mean ratio of hazard or progression rate of active treatment relative to placebo.

## 6.4 Interim Analysis

RGC will be considered for early stopping for futility according to the interim analysis schedule and definition specified in the "ALS Master Protocol Recommended Statistical Analysis, Design and Simulation Report" (Appendix 1 to the Master Protocol). RGC will not be stopped early for success.

## 6.5 Secondary Efficacy Analyses

#### 6.5.1 Hierarchical Testing

Primary inference for secondary efficacy endpoints will be based on analysis of the FAS analysis set using a joint-rank comparison for the combined assessment of function and survival (CAFS (Section 6.5.2 below), a repeated-measures linear mixed model for SVC (see Section 6.5.3 below), and Kaplan-Meier product-limit estimates and log-rank test for the primary survival endpoint (see Section 6.5.4 below) with a comparison between all active arm participants (i.e., the average of both 30 mg/d and 60 mg/d dosage groups) vs. placebo participants. The sequence for testing secondary efficacy endpoints is the following:

- 1. CAFS,
- 2. SVC,
- 3. Survival.

If the primary analysis indicates a significant slowing in disease progression from the Bayesian shared-parameter, repeated-measures model of ALSFRS-R and mortality, then each secondary efficacy endpoint in succession would be declared significant in the specified sequence using a comparison-wise criterion of two-tailed p < 0.05. After the first failure to declare significance, no endpoints lower in the hierarchy can be significant. This sequential closed-testing procedure controls the overall type 1 error rate at 5%. Nominal comparison-wise p-values for secondary efficacy endpoints will also be reported.

## 6.5.2 CAFS

The test consists of calculating a rank-sum score for each individual relative to pair-wise comparisons with all other participants. Participants are first ranked according to time to death or death equivalent when that is observed for both members of a pair or when one is censored after the observed event time for the other. Pairs that cannot be ranked by time to death or death equivalent are subsequently ranked by absolute change from baseline in ALSFRS-R total score at the maximum follow-up time at which both participants have an observation.

The primary CAFS analysis is the same as specified in the MPRDR with the clarification that the active treatment group pools participants randomized to 30 mg/d CNM-Au8 and 60 mg/d CNM-Au8.

The estimand is the stochastic probability that a randomly selected active participant will rank higher than a randomly selected placebo participant based on time to death or death equivalent or change from baseline in ALSFRS-R. The estimand is defined by the following attributes:

- Treatment: CNM-Au8 administered orally at dosages of 30 mg/d and 60 mg/d vs. placebo.
- Population: FAS population as defined in Section 6.1.
- Variables: ranksum for relative time to death or death equivalent up to the Week 24 Visit or absolute change from baseline in ALSFRS-R total score.
- Intercurrent event: treatment discontinuation: handled via treatment policy approach, with pair ranked comparisons up at the maximum follow-up time at which both participants have an observation.
- Population-level summary: difference in means of ranks of active treatment relative to placebo.

Inference from this analysis is supportive of inference from the Bayesian shared-parameter, repeated-measures model for the primary endpoint and is the primary analysis for this secondary endpoint.

The following SAS code specifies the analysis:

```
proc mixed data=work.cafs;
  class trtrnd(ref='0');
  model Rank = sx2bl dFRS rlz edv trtrnd / solution clparm;
  estimate "Active vs. Placebo (one-sided)" Treat 1 -1 / cl upper;
run;
```

where trtrnd indicates treatment group (active = 1 or placebo = 0), Rank is the sum of the ranks (-1, 0, 1) of each participant vs. every other participant in the FAS analysis set, sx2bl is years

since ALS symptom onset, dFRS is pre-baseline slope, rlz is an indicator of riluzole use at baseline, and edv is an indicator of edaravone use at baseline. A significant difference requires interpretation based on estimates from the survival analysis described in Section 6.5.4 and the repeated-measures analysis of ALSFRS-R total score described in Section 6.5.3.

In addition to the joint-rank CAFS analysis of PAV-free survival and change in ALSFRS-R total score including adjustment for covariates, the following additional joint-rank analyses will also be performed:

- 1. SVC will be analyzed as a joint-rank test by substituting the change from baseline of SVC in place of ALSFRS-R total score as an additional supportive analysis,
- 2. An additional set of joint-rank analyses will use multiple imputation to extend follow-up of (i) ALSFRS-R total score and (ii) SVC for participants who early terminate, withdraw consent, or are lost to follow-up as supportive analyses,
- 3. An additional set of joint-rank analyses for (i) ALSFRS-R total score and (ii) SVC will use time to death independent of any death equivalent as supportive analyses,
- 4. An additional set of joint-rank analyses for (i) ALSFRS-R total score and (ii) SVC will adjust rank scores in a linear model with the following covariates: time from ALS symptom onset, delta-FRS, baseline use of riluzole, baseline use of edaravone, and baseline serum NfL level, and
- 5. An additional set of joint-rank analyses for (i) ALSFRS-R total score and (ii) SVC without adjustment and comparing pairs of participants at the last jointly observed time point as sensitivity analyses.

The multiple imputation model referenced as method 2 above and used to extend follow-up of functional scores for participants who early terminate, withdraw consent, or are lost to follow-up will use linear regression with covariates of time since symptom onset, delta-FRS, baseline riluzole use, baseline edaravone use, and each observed functional score prior to a missing assessment.

Inference from the joint-rank analyses of SVC are supportive of inference from the repeated-measures model. Primary inference from the joint-rank CAFS analyses will compare survival by time to death or death equivalent, will compare change in function to the last jointly observed time point, and will adjust for the specified covariates.

#### 6.5.3 Repeated-measures Model

The specification of the repeated-measures linear mixed model and the primary linear contrast for estimating differences in 24-week change from baseline in a given continuous efficacy endpoint (ALSFRS-R total and domain scores, HHD upper extremity, lower extremity, and global average percentages, SVC, FVC by home spirometry, serum creatinine, serum NfL, urinary p75[ECD], ALSAQ-40 domain scores and SI, and CNS-BFS total score) are revised from those specified in the M-SAP to include a main effect of treatment and with the modification that treatment group is a three-level variable (i.e., placebo, 30 mg/d CNM-Au8, and 60 mg/d CNM-Au8).

The model will include fixed terms for discrete visit, treatment group (3 levels), treatment group × visit interaction, centered time since symptom onset × visit interaction, centered delta-FRS and centered delta-FRS × visit interaction, centered baseline riluzole use and centered baseline riluzole × visit interaction, and centered baseline edaravone

use and centered baseline edaravone × visit interaction. The following equations describe the model with regimen random effects:

$$Y_{ij} = a_{k(i)} + \gamma_1 t_i + \gamma_{2,j} v_j + \gamma_3' \mathbf{z}_i + \gamma_{4,j} t_i v_j + \gamma_{5,j}' \mathbf{z}_i v_j + \epsilon_{ij}$$

$$a_k \sim N(0, \sigma_r^2), \, \boldsymbol{\epsilon}_{i\cdot} \sim N(\mathbf{0}, \mathbf{R}), \, \text{Cov}(b_{k(i)}, \epsilon_{ij}) = 0$$
(eqn. 1)

where  $Y_{ij}$  is a given efficacy endpoint measured in participant i at visit j,  $a_{k(i)}$  is a random intercept for regimen k to which participant i was assigned,  $v_j$  is an indicator variable for visit j,  $z_i$  is the vector of covariates (centered time since onset, centered delta-FRS, centered baseline riluzole use, and centered baseline edaravone use) for participant i,  $t_i$  is an indicator variable for treatment t to which participant i was assigned,  $\gamma_l$ ,  $\gamma_{2,j}$ ,  $\gamma_3$ ,  $\gamma_{4,j}$ , and  $\gamma_{5,j}$  are estimated parameters and vectors of parameters for the fixed effects, and  $\epsilon_{ij}$  is the residual for participant i at visit j. The regimen-specific random effects are normally distributed with mean 0 and variance  $\sigma^2_r$ . The vector of residuals for a given participant are normally distributed with mean 0 and an unstructured covariance matrix  $\mathbf{R}$ . The regimen-specific random effect for a given participant and residuals for that participant are uncorrelated.

The following SAS code specifies the model:

where id is a participant study identifier, trtrnd is the randomly assigned treatment group, visit is the visit identifier, Value is value of the efficacy endpoint being tested for a given participant at a given visit, sx2b1 is years since ALS symptom onset centered at the sample median, dFRS is pre-baseline slope centered at the sample median, rlz is an indicator of riluzole use at baseline, and edv is an indicator of edaravone use at baseline. The primary estimate will be the treatment-dependent difference in change from baseline to the Week 24 Visit. The estimate and its 95% Wald confidence bounds will be obtained by a linear contrast of adjusted means.

The estimand estimated by the primary linear contrast of the shared-baseline, repeated-measures linear mixed model is the mean difference in 24-week change from baseline of a given continuous efficacy endpoint in the two active treatment groups relative to the placebo group in the FAS population. The estimand is defined by the following attributes:

- Treatment: CNM-Au8 administered orally at dosages of 30 mg/d and 60 mg/d vs. placebo.
- Population: FAS population as defined in Section 6.1.
- Variables: absolute change in endpoint from baseline to the Week 24 Visit.
- Intercurrent event: treatment discontinuation: handled via treatment policy approach, all data will be used including data collected during the placebo-controlled period after treatment discontinuation. Missing data post-treatment, including data missing due to death, will not be imputed, handled via missing at random assumption.

• Population-level summary: difference in conditional means of active treatment relative to placebo.

Inference from this analysis is supportive of inference from the Bayesian shared-parameter, repeated-measures model for the primary endpoint and is the primary analysis for the secondary SVC endpoint.

The following SAS code specifies the linear contrast for an endpoint measured every 8 weeks and assuming that the sort order for treatment group is placebo, 30 mg/d CNM-Au8, and 60 mg/d CNM-Au8 and visits are sorted chronologically:

```
estimate "3|Act vs Plb|dWk 24"
post*trtrnd*visit 2 0 0 -2 -1 0 0 1 -1 0 0 1 / cl divisor=2;
```

A significant difference in 24-week change in the direction of improved function would support inference that CNM-Au8 treatment reduced progression over 24 weeks for the efficacy endpoint being tested.

A separate supportive analysis for clinical endpoints (ALSFRS-R total and domain scores, HHD upper extremity, lower extremity, and global average percentages, SVC, FVC by home spirometry, ALSAQ-40 domain scores and SI, and CNS-BFS total score) will include centered baseline serum NfL level and the interaction of centered baseline serum NfL level and visit as additional covariates.

#### 6.5.4 Survival

The primary estimate of the effect of treatment on survival as an efficacy endpoint will include both death and death equivalent as components, will pool participants randomized to 30 mg/d CNM-Au8 and 60 mg/d CNM-Au8 in the FAS analysis set, and will include baseline age as an additional covariate in adjusted models. Otherwise, summaries and analyses of time to death or death equivalent are the same as specified in the M-SAP.

The estimand estimated by the logrank test is the deviation in expected survival times in the FAS population. The estimand is defined by the following attributes:

Treatment: CNM-Au8 administered orally at dosages of 30 mg/d and 60 mg/d vs. placebo.

Population: FAS population as defined in Section 6.1.

Variables: time to earlier of death or death equivalent.

Intercurrent event: treatment discontinuation: handled via treatment policy approach, all data will be used including data collected during the placebo-controlled period after treatment discontinuation. Missing data post-treatment will not be imputed, handled via missing completely at random assumption.

Population-level summary: difference in survival curves of active treatment and placebo.

In the presence of a significant different by the logrank test, inference on whether active treatment extended survival will be based on the hazard ratio estimated from an unadjusted Cox proportional hazards regression.

Survival to the end of the placebo-controlled period will also be analyzed in the ECM, ERO, EPP, STF, SFN, and SRO analysis sets. Survival analyses that include follow-up beyond the placebo-controlled period will be analyzed in the ERO analysis set.

Listings of all participants in the FAS, ECM, ERO, EPP, STF, and SRO analysis sets will document whether each participant had died, had reached a death equivalent endpoint, or was alive and free of a death equivalent and the study day of death, death equivalent, or last know alive and free of a death equivalent for each analysis timepoint.

## 6.5.5 Random-slopes Model

The specification of the random-slopes linear mixed model and the primary linear contrast for estimating differences in mean rate of progression in a given continuous efficacy endpoint (ALSFRS-R total and domain scores, HHD upper extremity, lower extremity, and global average percentages, SVC, FVC by home spirometry, quantitative voice characteristics, serum creatinine, serum NfL, urinary p75[ECD], ALSAQ-40 domain scores and SI, and CNS-BFS total score) are revised from those specified in the M-SAP to include a main effect of treatment and with the modification that treatment group is a three-level variable (i.e., placebo, 30 mg/d CNM-Au8, and 60 mg/d CNM-Au8).

The model will include fixed terms for month since the Baseline Visit, treatment group, treatment group × month interaction, centered years since ALS symptom onset and centered years since ALS symptom onset × month interaction, centered delta-FRS and centered delta-FRS × month interaction, centered baseline riluzole use and centered baseline riluzole use × month interaction, and centered baseline edaravone use and centered baseline edaravone use × month interaction. The following equations describe the model with regimen random effects:

$$Y_{ij} = \gamma_1 + a_{k(i)}^0 + b_i^0 + \gamma_2 t_i + \gamma_3' \mathbf{z}_i$$

$$+ \left(\gamma_4 + a_{k(i)}^1 + b_i^1 + \gamma_5 t_i + \gamma_6' \mathbf{z}_i\right) m_{ij} + \epsilon_{ij}$$

$$\{a_k^0, a_k^1\} \sim N(\mathbf{0}, \mathbf{\Sigma}_r), \{b_k^0, b_k^1\} \sim N(\mathbf{0}, \mathbf{\Sigma}_p), \epsilon_{ij} \sim N(\mathbf{0}, \sigma_\epsilon^2)$$

$$Cov(\mathbf{a}_k, \mathbf{b}_k) = \mathbf{0}, Cov(\mathbf{a}_k, \epsilon_{i\cdot}) = \mathbf{0}, and Cov(\mathbf{b}_k, \epsilon_{i\cdot}) = \mathbf{0}$$
(eqn. 2)

where  $Y_{ij}$  is a given efficacy endpoint measured in participant i at visit j,  $a^0_{k(i)}$  and  $a^1_{k(i)}$  are random intercept and slope for regimen k to which participant i was assigned,  $b^0_i$  and  $b^1_i$  are random intercept and slope for participant i,  $z_i$  is the vector of covariates (centered time since onset, centered delta-FRS, centered baseline riluzole use, and centered baseline edaravone use) for participant i,  $m_{ij}$  is the time from baseline to observation j for participant i in months calculated as days x 12 / 365.25,  $t_i$  is an indicator variable for treatment t to which participant i was assigned,  $\gamma_1$ ,  $\gamma_2$ ,  $\gamma_3$ ,  $\gamma_4$ ,  $\gamma_5$ , and  $\gamma_6$  are estimated parameters and vectors of parameters for the fixed effects, and  $\epsilon_{ij}$  is the residual for observation j for participant i. The regimen-specific random effects are normally distributed with mean  $\mathbf{0}$  and unstructured covariance matrix  $\mathbf{\Sigma}_r$ . The participant-specific random effects are normally distributed with mean  $\mathbf{0}$  and unstructured covariance matrix  $\mathbf{\Sigma}_p$ . The residuals for a given participant are normally distributed with mean  $\mathbf{0}$  and variance  $\sigma^2_{\epsilon}$ . The regimen-specific random effects, participant-specific random effects, and residuals are uncorrelated.

The following SAS code specifies the model:

```
random intercept month / subject=id type=un;
```

where month is time in months from the Baseline Visit (assuming 12 months in an average of 365.25 days per year) and other fields are the same as identified above in Section 6.5.3. The primary estimand will be the treatment-dependent difference in slopes. The estimate and its 95% Wald confidence bounds will be obtained by a linear contrast of adjusted means.

The estimand estimated by the primary linear contrast of the random-slopes linear mixed model is the difference in mean rate of progression of a given continuous efficacy endpoint in the two active treatment groups relative to the placebo group in the FAS population. The estimand is defined by the following attributes:

Treatment: CNM-Au8 administered orally at dosages of 30 mg/d and 60 mg/d vs. placebo.

Population: FAS population as defined in Section 6.1.

Variables: mean rate of change in endpoint from baseline to the Week 24 Visit.

Intercurrent event: treatment discontinuation: handled via treatment policy approach, all data will be used including data collected during the placebo-controlled period after treatment discontinuation. Missing data post-treatment will not be imputed, handled via missing at random assumption.

Population-level summary: difference in conditional mean slopes of active treatment relative to placebo.

Inference from these analyses is supportive of inference from the Bayesian shared-parameter, repeated-measures model for the primary endpoint and inference from the repeated-measures linear mixed model for secondary endpoints.

The following SAS code specifies the linear contrast assuming that the sort order for treatment group is placebo, 30 mg/d CNM-Au8, and 60 mg/d CNM-Au8:

A significant difference in slopes in the direction of improved function would support inference that the treatment reduced rate of progression for the efficacy endpoint being tested.

A separate supportive analysis for clinical endpoints (ALSFRS-R total and domain scores, HHD upper extremity, lower extremity, and global average percentages, SVC, FVC by home spirometry, quantitative voice characteristics, ALSAQ-40 domain scores and SI, and CNS-BFS total score) will include centered baseline serum NfL level and the interaction of centered baseline serum NfL level and study month as additional covariates.

## **6.5.6** Time to Clinical Events

Time to hospitalizations and clinical events will be analyzed in the FAS, ECM, ERO, and EPP analysis sets. The summaries and analyses will parallel the analyses described for survival described in Section 6.5.4. Analysis of time to King's stage 4a or 4b and time to a 6-point decline in ALSFRS-R total score will accommodate interval censoring between ALSFRS-R assessments. Analysis of time to King's stage 4a or 4b will be stratified by baseline King's stage.

## 6.5.7 Composite of ALSFRS-R, SVC, and ALSAQ-40 Slopes

Participant-specific rates of change in ALSFRS-R total score, SVC percent-predicted, and ALSAQ-40 total score will be estimated in separate, endpoint-specific unadjusted random-slopes linear mixed models in the FAS, ECM, and ERO analysis sets. Participant-specific random slopes for each endpoint will be standardized to a mean of zero (0) and a variance of one (1) and then averaged for each participant. The composite average of standardized random slope estimates will be compared across treatment groups by one-way analysis of variance with adjustment for the following median-centered covariates: years since ALS symptom onset, delta-FRS, baseline riluzole use, and baseline edaravone use. A separate analysis will include baseline serum NfL level as an additional covariate. Treatment comparison between all active arm participants (i.e., the average of both 30 mg/d and 60 mg/d dosage groups) vs. placebo participants and between each active treatment group separate vs. placebo will be estimated using contrasts of least-square means.

## 6.5.8 HHD0 and HHD0<sup>2</sup>

Analyses of HHD0 are the same as specified in the M-SAP with the modification that treatment group is a three-level variable (i.e., placebo, 30 mg/d CNM-Au8, and 60 mg/d CNM-Au8), with addition of parallel analyses of HHD0<sup>2</sup>, with a separate analysis that includes baseline serum NfL level as an additional covariate, and with the clarification that time to zero strength for both analyses is interval censored between HHD assessments.

Inference from these analyses is supportive of inference from the repeated-measures linear mixed model for HHD upper and lower extremity scores.

#### **6.5.9 Quantitative Voice Measures**

Given the high frequency of voice recordings, a repeated-measures analysis with unstructured covariance is overly flexible but the assumption of linear change required by the random-slopes model may be overly rigid. To complement estimates from the random-slopes linear mixed model, quantitative voice characteristics will be analyzed in a linear mixed model in which the temporal profile for both fixed and random terms is modeled using cubic B-splines with knots at 8 and 16 weeks. The model will include fixed terms for B-splines (4 terms), treatment group (3 levels), treatment group × B-spline interaction, centered time since symptom onset and centered time since symptom onset × B-spline interaction, centered delta-FRS and centered delta-FRS × B-spline interaction, centered baseline riluzole use and centered baseline riluzole × B-spline interaction, and centered baseline edaravone use and centered baseline edaravone × B-spline interaction. The model will include random regimen-specific intercepts and slopes with unstructured covariance, random participant-specific B-splines (5 terms) with unstructured covariance, and a first-order autoregressive structure for residuals. A simplified covariance structure assuming no regimen-level covariance, heterogeneous compound symmetric covariance among the random B-splines, conditional independence of residuals, or a combination of the three simplifying assumptions will be used if the full model fails to converge. The primary estimand will be the active (i.e., the average of both 30 mg/d and 60 mg/d dosage groups) vs. placebo treatment-dependent difference in 24-week change from baseline. The estimate and its 95% Wald confidence bounds will be obtained by a linear contrast of adjusted means.

A separate supportive analysis will include centered baseline serum NfL level and the interaction of centered baseline serum NfL level and B-splines as additional covariates.

## 6.5.10 Placebo Multiple Imputation

Placebo multiple imputation analyses are the same as specified in the M-SAP with the modification that treatment group is a three-level variable (i.e., placebo, 30 mg/d CNM-Au8, and 60 mg/d CNM-Au8). Placebo multiple imputation analyses will be applied to ALSFRS-R total score, HHD upper and lower extremity percentages, and SVC.

The following SAS code specifies the imputation for an endpoint measured every 8 weeks:

where Wk00, Wk08, Wk16, and Wk24 are the values of a given efficacy endpoint at the Baseline, Week 8, Week 16, and Week 24 Visits, respectively, trtnd has a value of zero (0) for participants randomized to placebo, and x and y take appropriate values to specify the range of a given outcome measure (i.e., 0 and 48 for ALSFRS-R total score; 0 and . for HHD upper and lower extremity percentages and SVC).

Inference from these analyses is supportive of inference from the Bayesian shared-parameter, repeated-measures model for the primary endpoint and assess sensitivity to the missing data assumption of the repeated-measures linear mixed model for secondary endpoints in the FAS analysis set. A separate analysis will include centered baseline serum NfL level as an additional covariate in both imputation stages.

## 6.5.11 Additional Sensitivity Analyses of Primary and Key Secondary Outcomes

Sensitivity analyses of primary and key secondary efficacy outcomes are the same as specified in the M-SAP with the modification that treatment group is a three-level variable (i.e., placebo, 30 mg/d CNM-Au8, and 60 mg/d CNM-Au8).

#### **6.5.12 Subgroup Analyses**

In addition to the subgroups specified in the M-SAP, the following additional subgroups will be analyzed in the random-slope model (see Section 6.5.5) for primary and secondary efficacy endpoints in the FAS analysis set:

- Baseline use of riluzole and edaravone (neither, riluzole only, edaravone only, both),
- Age (less than 65 years vs. 65 years or older),
- Sex (female vs. male),
- Race (white vs. any minority race with greater than 5% prevalence in the sample),
- Ethnicity (Hispanic or Latino vs. non-Hispanic or Latino),

- Weight (less than 43 kg, 43 to less than 56 kg, 56 to less than 77 kg, 77 to less than 150 kg, 150 kg or more),
- BMI (less than  $18.5 \text{ kg/m}^2$ ,  $18.5 \text{ to less than } 25 \text{ kg/m}^2$ ,  $25 \text{ to less than } 30 \text{ kg/m}^2$ ,  $30 \text{ to less than } 40 \text{ kg/m}^2$ ,  $40 \text{ kg/m}^2$  or more),
- Chronic kidney disease (CKD) stage (stage 1 or better [eGFR 90 mL/min/1.73m<sup>2</sup> or more], stage 2 [eGFR 60 to 89 mL/min/1.73m<sup>2</sup>], stage 3 [eGFR 30 to 59 mL/min/1.73m<sup>2</sup>], stage 4 [eGFR 15 to 29 mL/min/1.73m<sup>2</sup>], stage 5 [eGFR less than 15 mL/min/1.73m<sup>2</sup>]),
- Time since onset of weakness (less than 18 months vs. 18 months or longer),
- El Escorial and time since onset of weakness (El Escorial definite and less than 18 months vs. not both),
- Baseline symptom severity (all ALSFRS-R questions scored 2 or greater vs. any question scored 0 or 1),
- Early disease state (all ALSFRS-R questions scored 2 or greater, SVC 80%-predicted or greater, and time since symptom onset less than 24 months vs. not meeting all three criteria),
- Baseline serum urate concentration (less than 5.5 mg/dL vs. 5.5 mg/dL or greater),
- Baseline serum NfL concentration (by median split),
- Baseline delta-FRS score (less than 0.47 points/year, 0.47 to less than 1.11 points/year, 1.11 points/year or greater),
- Site of onset (any bulbar onset, no bulbar onset),
- Site (individual sites with at least 5 participants per treatment group and all participants from sites with fewer than 5 participants per treatment group pooled).

For each classification, unknown, not reported, and missing will be considered one group. All individuals not included in a specified subgroup will be combined into a mixed, "other" group. The "other" group will be included in analyses if its prevalence is greater than 5%; otherwise, the "other" group will be excluded.

In cases where a model for a given subgroup and endpoint fails to converge, the covariance terms for the regimen-specific random effects will be simplified from unstructured covariance of intercepts and slopes to separate, uncorrelated variance components for intercepts and slopes. If convergence still fails, regimen-specific intercepts and slopes will be modeled as fixed effects. If convergence still fails, the participant-specific random effects will be simplified from unstructured covariance of intercepts and slopes to separate, uncorrelated variance components for intercepts and slopes.

#### 6.5.13 Comparison of Controls across Regimens

Comparisons of placebo participants across regimens are the same as specified in the M-SAP with separate analyses that include baseline serum NfL level as an additional covariate plus applicable interaction terms as relevant to a given model.

## 6.5.14 Pharmacokinetic Analyses of CNM-Au8

Pre-dose concentrations of CNM-Au8 in whole blood and plasma will be summarized by treatment group and visit in the ERO sample. Concentrations below the limit of quantitation (BLQ) will be replaced with one half of the lower limit of quantitation. Summaries will include number of observations, number and percentage with concentrations BLQ, arithmetic mean, median, standard deviation, minimum, maximum, geometric mean, geometric coefficient of variation (calculated as sqrt(exp(variance of log-transformed concentrations) – 1)), and 95% confidence bounds for the geometric mean assuming log-normally distributed data.

A concentration response relationship based on observed CNM-Au8 C<sub>max</sub> per active participant versus ALSFRS-R slope change will also be analyzed as an exploratory endpoint.

Whole blood and plasma concentration data of CNM-Au8 may be subjected to population pharmacokinetic analysis to derive population estimates of pharmacokinetic parameters and test the effect of various covariates such as age, weight, and sex. Details of the analysis will be described in a separate data analysis plan (DAP). This analysis may be performed by combining data from the current study with data from other studies of CNM-Au8, if deemed appropriate. The tests of association with ALSFRS-R and the population pharmacokinetic analysis will be performed by Clene Nanomedicine or its designee and reported in a separate modelling report.

## 6.5.15 Pharmacodynamic Biomarker Analyses

Pharmacodynamic biomarkers other than serum creatinine, serum and CSF NfL, and urinary p75[ECD] will be analyzed by Clene Nanomedicine according to a separate pharmacodynamic DAP (Regimen C Pharmacodynamic Analysis Plan) and will be reported in a separate report.

#### 6.5.16 Pharmacokinetics of Riluzole

Pharmacokinetic analysis of plasma riluzole concentrations will be analyzed according to a separate pharmacokinetic analysis plan authored and conducted by Dr. Charles Venuto, PharmD.

#### 6.6 Safety Analyses

## **6.6.1** Treatment-emergent Adverse Events

Summaries and analyses of treatment-emergent adverse events (TEAE) are the same as specified in the M-SAP with the following revisions.

TEAEs are defined as those adverse events with onset dates in the interval from double-blind treatment initiation to either the Final Safety Visit if completed, the date of death if the participant dies, 28 days after last dose of study drug if the participant early terminates or is lost to follow-up, or the date of first dose of study drug during participation in the OLE, if so exposed. Adverse events with onset on the day of double-blind treatment initiation and adverse events with incompletely specified onset date where the ambiguous date spans the day of double-blind treatment initiation will be assumed to be treatment emergent except for those known to precede first exposure to study drug.

In addition to summaries specified in the M-SAP, serious TEAEs will be summarized by MedDRA system organ class, high level term, and preferred term for all TEAEs. In addition, TEAEs will be summarized by Medical Dictionary for Regulatory Activities (MedDRA) system organ class and preferred term for fatal TEAEs, TEAEs that occurred during a participant's COVID-19 infection (defined as 5 days prior to symptom onset to end of COVID-19 symptoms


or the earlier of 91 days after symptom onset or the end of double-blind follow-up, if ongoing), and TEAEs and serious TEAEs stratified by the following subgroups: baseline riluzole use, baseline edaravone use, age, sex, race, ethnicity, weight, BMI, and CKD stage. Subgroup classifications will be the same as described in Section 6.5.12 Subgroup Analyses except that the "other" group will be retained regardless of prevalence.

TEAEs indicating COVID-19 infection are the following: Asymptomatic COVID-19, COVID-19, COVID-19 pneumonia, COVID-19 treatment, Post-acute COVID-19 syndrome, SARS-CoV-2 antibody test positive, SARS-CoV-2 RNA increased, SARS-CoV-2 sepsis, SARS-CoV-2 test false negative, SARS-CoV-2 test positive, SARS-CoV-2 viraemia, Suspected COVID-19.

Treatment-dependent differences in the proportion of participants experiencing a given type of TEAE will not be tested. Treatment-dependent differences in TEAE incidence rates in units of number per 100 participant years will be estimated as differences rather than ratios and will include comparison-wise 95% confidence intervals with variance estimates obtained by the delta method.

## 6.6.2 Safety Labs

Summaries and analyses of clinical safety labs are the same as specified in the M-SAP with the revision that abnormal levels will be classified to a toxicity grade based on quantitative grading using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 and with the addition that maximum toxicity over all post-baseline visits will be included in shift tables along with visit-specific shifts.

The proportion of participants with ALT >3x ULN, AST >3x ULN, creatinine >1.5x level at the Baseline Visit, and platelet count <75,000/mm³, or with any of the four will be presented as shift tables vs. the status of each participant at baseline for each visit by treatment group in all safety samples. The absolute level and the absolute change from baseline for ALT, AST, creatinine, and platelet count will be summarized as means, standard deviations, medians, and ranges at each visit by treatment group in all safety samples.

#### 6.6.3 ECG Results

Summaries of ECG parameters and findings are the same as specified in the M-SAP.

#### 6.6.4 Vital Signs and Weight

Summaries and analyses of vital signs and weight are the same as specified in the M-SAP.

#### 6.6.5 Suicidality

Summaries of suicidality are the same as specified in the M-SAP.

## 6.7 Other Analyses

## 6.7.1 Participant Disposition

All participants consented to the Master Protocol between the time of the first and last consent of a participant assigned to a regimen included in the FAS analysis set will be summarized as a single set for the following events: consented to the Master Protocol, failed screening for the Master Protocol, other reasons not assigned to a regimen (including timing out of the screening window, death, withdrawal of consent, early termination, and administrative termination), and assigned to a regimen. Reasons for Master Protocol screen failure will be summarized.


All participants in the above sample assigned to a regimen will be summarized as two sets (final screening for RGC vs. final screening for a non-RGC regimen) for the following events: consented to a regimen, failed screening for a regimen, other reasons not randomized within a regimen (including timing out of the screening window, death, withdrawal of consent, early termination, and administrative termination), and randomized within a regimen. If a given individual is screened multiple times prior to randomization within a regimen, then the final screening experience of that individual will be summarized. Reasons for RGC screen failure will be summarized separately for all participants screened for RGC whether that was their final screening experience or not.

All participants in the FAS analysis set will be summarized as two sets (randomization to active study drug vs. randomization to placebo) for the following events: initiated regimen-specific study drug, prematurely terminated study participation due to death, withdrawal of consent, early termination, loss to follow-up, or administrative termination, completed 24-week follow up, and completed a safety follow-up visit vs. continued into the OLE. Reasons for withdrawal of consent or early termination after randomization will be summarized.

Any randomized participants excluded from the FAS and EPP analysis sets or included in the FAS analysis set but not contributing to the primary analysis will be identified in a listing together with the reason for their exclusion.

## 6.7.2 Study Drug Compliance and Tolerance

Summaries of study drug compliance and tolerance are the same as specified in the M-SAP with the clarification that summaries will be reported for the ERO and SRO analysis sets and that date of permanent discontinuation of study drug is the date of last use of double-blind study drug among all participants in a given analysis set.

The number of days of exposure to study drug will be calculated in three ways:

- as the number of days from dose initiation to the final safety assessment during the placebocontrolled period, inclusive,
- as the number of days from dose initiation to drug withdrawal, inclusive, less any interval during which use of study drug was interrupted (individual missed doses will not be subtracted unless noted in the dosage management log), and
- as the number of days from dose initiation to the earlier of final contact during the placebocontrolled period or 28 days after last dose of study drug, inclusive.

The proportion of participants who interrupted study drug or reduced study drug dosage and the time to first study drug interruption or dosage reduction will be summarized. The number of days of exposure to a reduced dosage of study drug will be summarized.

#### 6.7.3 Concomitant Medication Use

Summaries of concomitant medication use are the same as specified in the M-SAP with the clarification that medications taken at baseline and those initiated after first dose of study drug will be separately summarized and will be classified by ATC Therapeutic class and WHODrug Preferred base name.

#### 6.7.4 Medical History

Medical histories will be summarized by MedDRA system organ class, high level term, and preferred term in the STF and SRO analysis sets.

#### 6.7.5 Blindedness

The proportions of participants and site investigators who report on the Exit Questionnaire a guess of active vs. placebo treatment assignment, each level of surety of that guess, and each of five pre-specified reasons for making a treatment assignment will be summarized by treatment group in the FAS and ERO analysis sets. Treatment-dependent differences in the proportion guessing active treatment assignment will be tested among all respondents and among those stating they are at least somewhat sure of their guess by Fisher's exact test and the difference in proportion guessing active treatment assignment will be estimated with confidence bounds.

#### 6.7.6 Protocol Deviations

The number of major and minor protocol deviations will be summarized by type of deviation and treatment group in all analysis sets. Listings of all protocol deviations will be produced.

## 6.7.7 Impact of COVID-19 Pandemic

The proportions of planned assessments missed due to COVID-19 restrictions or disruptions will be summarized by treatment group, visit, and type of assessment in the FAS and ERO analysis sets. Protocol deviations that resulted from COVID-19 restrictions or disruptions will be summarized by treatment group and type of deviation in the FAS and ERO analysis sets and listed.

#### 7. Validation

## 7.1 Primary Efficacy Analysis

Validation of the primary efficacy analysis is the same as specified in the M-SAP.

## 7.2 Secondary, Exploratory, and Safety Analyses

Validation of secondary, exploratory, and safety analyses are the same as specified in the M-SAP.

#### 8. References

The following references are cited in addition to those specified in the M-SAP:

Balendra R, Jones A, Jivraj N, Knights C, Ellis CM, Burman R, Turner MR, Leigh PN, Shaw CE, Al-Chalabi A. Estimating clinical stage of amyotrophic lateral sclerosis from the ALS Functional Rating Scale. Amyotroph Lateral Scler Frontotemporal Degener. 2014 Jun;15(3-4):279-84.

Roche JC, Rojas-Garcia R, Scott KM, Scotton W, Ellis CE, Burman R, Wijesekera L, Turner MR, Leigh PN, Shaw CE, Al-Chalabi A. A proposed staging system for amyotrophic lateral sclerosis. Brain. 2012 Mar;135(Pt 3):847-52.


# **DocuSign**

#### **Certificate Of Completion**

Envelope Id: ACA6427AFF8F4849ACD6646E87B8086A

Subject: Please DocuSign: HEALEY ALS Platform RGC R-SAP v3.0 20220722\_unsigned.pdf

Source Envelope:

Document Pages: 37 Certificate Pages: 6

AutoNav: Enabled

**Envelopeld Stamping: Disabled** 

Time Zone: (UTC-05:00) Eastern Time (US & Canada)

Status: Completed

Envelope Originator: Marianne Chase

mchase@mgh.harvard.edu IP Address: 73.60.69.9

Sent: 7/22/2022 7:04:17 PM

Sent: 7/22/2022 7:04:18 PM

Viewed: 7/22/2022 7:05:40 PM

Signed: 7/22/2022 7:06:12 PM

Viewed: 7/23/2022 12:53:42 PM

Signed: 7/23/2022 12:54:49 PM

## **Record Tracking**

Status: Original

7/22/2022 7:00:35 PM

Holder: Marianne Chase

mchase@mgh.harvard.edu

Location: DocuSign

**Timestamp** 

## **Signer Events**

Ben Saville

ben@berryconsultants.net

Ben Saville

Security Level: Email, Account Authentication

(Required), Logged in

tion

Signature Adoption: Pre-selected Style

Signature ID:

**Signature** 

Ben Saville

Signatures: 6

Initials: 0

50221BD2-F3C9-432B-9863-2C6FEC7283AD

Using IP Address: 107.115.5.95

With Signing Authentication via DocuSign password

With Signing Reasons (on each tab):

I approve this document

## Electronic Record and Signature Disclosure:

Accepted: 6/24/2020 5:24:44 PM

ID: 0826203a-7d83-4395-a4f0-c1a7f44f1ee4

Eric A. Macklin

emacklin@mgh.harvard.edu

Instructor in Medicine

Eric Macklin

Security Level: Email, Account Authentication

(Required)

Eric A. Macklin

Signature Adoption: Pre-selected Style

Signature ID:

8E847DD4-0E85-42A1-B334-DFC089673751

Using IP Address: 173.48.212.201

With Signing Authentication via DocuSign password

With Signing Reasons (on each tab):

I approve this document

#### **Electronic Record and Signature Disclosure:**

Accepted: 5/8/2020 9:17:52 AM

ID: 2308ba7c-abcd-4949-872e-021ea95dc489

| Signer Events | Signature | Timestamp |
|---|---|---|
| Merit Cudkowicz<br>cudkowicz.merit@mgh.harvard.edu<br>Chief of Neurology | Merit Cudkowicz | Sent: 7/22/2022 7:04:19 PM<br>Viewed: 7/22/2022 7:21:00 PM<br>Signed: 7/22/2022 7:21:15 PM |
| Security Level: Email, Account Authentication (Required) | Signature Adoption: Pre-selected Style Signature ID: 9F8FE418-0E50-4C6A-B0A6-7B835E80C644 Using IP Address: 108.26.176.128 | |
| | With Signing Authentication via DocuSign password With Signing Reasons (on each tab): | |
| Electronic Record and Signature Disclosure:<br>Accepted: 7/22/2022 7:21:00 PM<br>ID: dcb30df1-d809-41d9-9561-b5a072bf1c47 | I approve this document | |
| Michael Hotchkin<br>michael.hotchkin@clene.com<br>Chief Development Officer | Michael Hotchkin | Sent: 7/22/2022 7:04:20 PM<br>Viewed: 7/22/2022 7:08:19 PM<br>Signed: 7/22/2022 7:08:42 PM |
| Clene Nanomedicine Inc. | | 0.9.104. 1,22,2022 1.001.2 1.11 |
| Security Level: Email, Account Authentication (Required) | Signature Adoption: Pre-selected Style Signature ID: | |
| | 1EBE8E10-E772-4615-A382-BBAE79F936CA<br>Using IP Address: 50.255.193.14 | |
| | With Signing Authentication via DocuSign password With Signing Reasons (on each tab): I approve this document | |
| Electronic Record and Signature Disclosure:<br>Accepted: 3/18/2022 10:04:00 AM<br>ID: 7797c6a2-b232-47fc-a9d6-5d05a268d034 | • | |
| Robert Glanzman | ٠, | Sent: 7/22/2022 7:04:19 PM |
| Robert@clene.com | d7- | Viewed: 7/22/2022 8:05:44 PM |
| Chief Medical Officer | , | Signed: 7/22/2022 8:06:29 PM |
| Security Level: Email, Account Authentication (Required) | Signature Adoption: Drawn on Device Signature ID: | |
| | D169CA24-5CAF-4E74-982A-7D386FF9400C | |
| | Using IP Address: 136.36.241.79 | |
| | Signed using mobile | |
| | With Signing Authentication via DocuSign password | |
| | With Signing Reasons (on each tab): I approve this document | |
| Electronic Record and Signature Disclosure:<br>Accepted: 7/22/2022 8:05:44 PM<br>ID: 1752ba69-ff7c-44a6-b1a9-1d45cb123774 | •• | |

**Signer Events** Sabrina Paganoni

Spaganoni@mgh.harvard.edu MD PhD

MGH

Security Level: Email, Account Authentication (Required)

**Signature** 

—DocuSigned by Sabrina Paganoni Sabrina Paganoni

**Timestamp** 

Sent: 7/22/2022 7:04:20 PM

Viewed: 7/22/2022 8:34:40 PM

Signed: 7/22/2022 8:35:04 PM

| I approve this document | 07/22/2022 | 5:35:01 PM PDT

-58705BF61CB842A887521BEB826294FA

Signature Adoption: Pre-selected Style

Signature ID:

58705BF6-1CB8-42A8-8752-1BEB826294FA

Using IP Address: 73.182.245.163

With Signing Authentication via DocuSign password

With Signing Reasons (on each tab):

I approve this document

**Electronic Record and Signature Disclosure:** 

Accepted: 7/22/2022 8:34:40 PM

ID: c9dcf81b-ce13-4b7a-8f17-ddc4960d0b47

| In Person Signer Events | Signature | Timestamp |
|---|---|---|
| Editor Delivery Events | Status | Timestamp |
| Agent Delivery Events | Status | Timestamp |
| Intermediary Delivery Events | Status | Timestamp |
| Certified Delivery Events | Status | Timestamp |
| Carbon Copy Events | Status | Timestamp |
| Witness Events | Signature | Timestamp |
| Notary Events | Signature | Timestamp |
| Envelope Summary Events | Status | Timestamps |
| Envelope Sent Certified Delivered Signing Complete Completed | Hashed/Encrypted Security Checked Security Checked Security Checked | 7/22/2022 7:04:20 PM<br>7/22/2022 8:34:40 PM<br>7/22/2022 8:35:04 PM<br>7/23/2022 12:54:49 PM |
| Payment Events | Status | Timestamps |
| Electronic Record and Signature Disclosure | | |

## ELECTRONIC RECORD AND SIGNATURE DISCLOSURE

From time to time, Insight OBO The Massachusetts General Hospital (we, us or Company) may be required by law to provide to you certain written notices or disclosures. Described below are the terms and conditions for providing to you such notices and disclosures electronically through the DocuSign system. Please read the information below carefully and thoroughly, and if you can access this information electronically to your satisfaction and agree to this Electronic Record and Signature Disclosure (ERSD), please confirm your agreement by selecting the check-box next to 'I agree to use electronic records and signatures' before clicking 'CONTINUE' within the DocuSign system.

# Getting paper copies

At any time, you may request from us a paper copy of any record provided or made available electronically to you by us. You will have the ability to download and print documents we send to you through the DocuSign system during and immediately after the signing session and, if you elect to create a DocuSign account, you may access the documents for a limited period of time (usually 30 days) after such documents are first sent to you. After such time, if you wish for us to send you paper copies of any such documents from our office to you, you will be charged a \$0.00 per-page fee. You may request delivery of such paper copies from us by following the procedure described below.

#### Withdrawing your consent

If you decide to receive notices and disclosures from us electronically, you may at any time change your mind and tell us that thereafter you want to receive required notices and disclosures only in paper format. How you must inform us of your decision to receive future notices and disclosure in paper format and withdraw your consent to receive notices and disclosures electronically is described below.

#### Consequences of changing your mind

If you elect to receive required notices and disclosures only in paper format, it will slow the speed at which we can complete certain steps in transactions with you and delivering services to you because we will need first to send the required notices or disclosures to you in paper format, and then wait until we receive back from you your acknowledgment of your receipt of such paper notices or disclosures. Further, you will no longer be able to use the DocuSign system to receive required notices and consents electronically from us or to sign electronically documents from us

## All notices and disclosures will be sent to you electronically

Unless you tell us otherwise in accordance with the procedures described herein, we will provide electronically to you through the DocuSign system all required notices, disclosures, authorizations, acknowledgements, and other documents that are required to be provided or made available to you during the course of our relationship with you. To reduce the chance of you inadvertently not receiving any notice or disclosure, we prefer to provide all of the required notices and disclosures to you by the same method and to the same address that you have given us. Thus, you can receive all the disclosures and notices electronically or in paper format through the paper mail delivery system. If you do not agree with this process, please let us know as described below. Please also see the paragraph immediately above that describes the consequences of your electing not to receive delivery of the notices and disclosures electronically from us.

## How to contact Insight OBO The Massachusetts General Hospital:

You may contact us to let us know of your changes as to how we may contact you electronically, to request paper copies of certain information from us, and to withdraw your prior consent to receive notices and disclosures electronically as follows:

To contact us by email send messages to: jhenrique@mgh.harvard.edu

## To advise Insight OBO The Massachusetts General Hospital of your new email address

To let us know of a change in your email address where we should send notices and disclosures electronically to you, you must send an email message to us at jhenrique@mgh.harvard.edu and in the body of such request you must state: your previous email address, your new email address. We do not require any other information from you to change your email address.

If you created a DocuSign account, you may update it with your new email address through your account preferences.

## To request paper copies from Insight OBO The Massachusetts General Hospital

To request delivery from us of paper copies of the notices and disclosures previously provided by us to you electronically, you must send us an email to jhenrique@mgh.harvard.edu and in the body of such request you must state your email address, full name, mailing address, and telephone number. We will bill you for any fees at that time, if any.

# To withdraw your consent with Insight OBO The Massachusetts General Hospital

To inform us that you no longer wish to receive future notices and disclosures in electronic format you may:

i. decline to sign a document from within your signing session, and on the subsequent page, select the check-box indicating you wish to withdraw your consent, or you may;

ii. send us an email to jhenrique@mgh.harvard.edu and in the body of such request you must state your email, full name, mailing address, and telephone number. We do not need any other information from you to withdraw consent.. The consequences of your withdrawing consent for online documents will be that transactions may take a longer time to process..

## Required hardware and software

The minimum system requirements for using the DocuSign system may change over time. The current system requirements are found here: <a href="https://support.docusign.com/guides/signer-guide-signing-system-requirements">https://support.docusign.com/guides/signer-guide-signing-system-requirements</a>.

## Acknowledging your access and consent to receive and sign documents electronically

To confirm to us that you can access this information electronically, which will be similar to other electronic notices and disclosures that we will provide to you, please confirm that you have read this ERSD, and (i) that you are able to print on paper or electronically save this ERSD for your future reference and access; or (ii) that you are able to email this ERSD to an email address where you will be able to print on paper or save it for your future reference and access. Further, if you consent to receiving notices and disclosures exclusively in electronic format as described herein, then select the check-box next to 'I agree to use electronic records and signatures' before clicking 'CONTINUE' within the DocuSign system.

By selecting the check-box next to 'I agree to use electronic records and signatures', you confirm that:

- You can access and read this Electronic Record and Signature Disclosure; and
- You can print on paper this Electronic Record and Signature Disclosure, or save or send this Electronic Record and Disclosure to a location where you can print it, for future reference and access; and
- Until or unless you notify Insight OBO The Massachusetts General Hospital as described above, you consent to receive exclusively through electronic means all notices, disclosures, authorizations, acknowledgements, and other documents that are required to be provided or made available to you by Insight OBO The Massachusetts General Hospital during the course of your relationship with Insight OBO The Massachusetts General Hospital.